CLINICAL TRIAL: NCT02432989
Title: Rest vs. Early Return to Exercise Following Concussion (H15-00307)
Brief Title: Establishing Early Exercise Interventions in Concussion Recovery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to get enough participants
Sponsor: University of British Columbia (Other)
Collaborators: Fortius Sport & Health (Other)
Responsible Party: Principal Investigator, Naznin Virji-Babul, Dr. Naznin Virji-Babul, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H15-00307
Record Dates: First submitted 2015-03-26; First posted 2015-05-04 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-03

CONDITIONS: Brain Concussion
Keywords: Exercise Therapy; Concussion Management; Concussion Recovery
MeSH Terms: conditions — Brain Concussion | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resting Control Group (No Intervention): Patients will receive standard concussion management, but will be asked not to exercise for the first 7 days after their concussion.
- Exercise Group (Experimental): Patients will receive standard concussion management, but will be asked to exercise on a stationary bike on two different occasions (once for 15 minutes and again for 30 minutes) in their first week of recovery. This group will also be asked to complete a 30 minute leisurely walk at their convenience on the two days they are not tested at UBC or Fortius.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Light-moderate exercise on a stationary bike and leisurely walks.
  Arms: Exercise Group

SUMMARY:
This is a Phase 1 study to determine (1) the safety of an exercise protocol in adolescents and young adults with concussion in the first week post-injury and (2) to evaluate the effects of mild symptoms on brain function using EEG. This pilot study will inform subsequent grant applications, and a Phase II randomized control trial that will explore the influence of age on an early re-introduction to exercise, as well as the influence of varying intensity levels of exercise.

DETAILED DESCRIPTION:
The investigators will recruit a total of 20 patients between the ages of 15-25.Ten patients will be randomized to the "rest" group and ten to the "exercise" group.

All patients will then be invited to complete balance testing and a 5 minute resting state EEG at the Perception Action Lab at UBC's Djavad Mowafaghian Centre for Brain Health within 48 hours of their concussion. At this time all patients will be provided with an Actigraph GT3X+ from Actigraph Corp and requested to wear this on their wrist or ankle 24 hours a day, and record times in which the device is removed. The patients will wear this device until returning to UBC on day 7 post-injury. Daily questionnaires describing their physical and mental activity levels, and any concussion related symptoms they experienced will also be completed. This initial meeting will take approximately 90 minutes.

Afterwards, all patients will be invited to attend a standard post-concussion management visit with a physical therapist at FORTIUS Sport and Health in Burnaby BC, 48-72 hours after their injury. Both the rest and exercise groups will receive a "standard post-concussion management visit". In this visit, physical measures of c-spine range of motion (ROM), c-spine proprioception with laser (within 7 cm pass, >7 cm fail), strength, presence/absence of subjective symptoms, numeric c-spine rating scale, and neurocognitive testing will be completed. Those assigned to the exercise group will additionally complete 15 minutes of light-moderate aerobic exercise on a stationary bike. Activity levels will be determined by the physical therapist to individualize each program using heart rate reserve (HHR) and perceived exertion between 11-12 on the Visual Analogue Scale (VAS) for "Rating of Perceived Exertion". Patients will aim to achieve 65% of their HHR. The visit will take approximately 60 minutes, with an additional 20 minutes for those assigned to the exercise group.

On day 4 post-injury, all patients will continue with the standard care and recovery at home, completing their daily questionnaires of activity levels and post-concussion symptom reporting. Those assigned to the exercise group will be asked to complete 30 minutes of continuous leisurely walking at their convenience.

All patients will complete a second standard post-concussion management visit to FORTIUS Sport and Health on day 5 or 6 post-injury to repeat their standard concussion care and neurocognitive testing. Those in the exercise group will be invited to complete 30 minutes of light-moderate aerobic exercise (65% HHR) on the stationary bike following the aforementioned criteria. On the remaining day, all patients will continue with standard care and recovery at home; completing their daily questionnaires of activity levels and post-concussion symptom reporting. Those in the exercise group will again complete 30 minutes of continuous leisurely walking at their convenience while at home.

On day 7 post-injury, patients will return to UBC for a follow up appointment in which balance testing, and resting state EEG will be re-assessed. Patients will return their Actigraph, and complete a final questionnaire. At this stage, participation will be considered complete

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in participating minor sports association in the Greater Vancouver Area
* Sustained a recent sports related concussion (within 48 hours of contacting the research coordinators)

Exclusion Criteria:

* Less than 15 years of age or over 25 years old.
* Diagnosis of concurrent learning disability, ADHD, Autism or Seizure.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in EEG Functional Connectivity Using Graph Theoretical Modeling | Within 48 hours of concussion, and 7 days post-injury
  Compare 5 minute resting state electroencephalogram (EEG) between rest and exercise groups. We will record the electrical activity (in Hertz) and compare values using Graph Theoretical measures that establish both global and local connectivity. We will look at the changes in composite measures of betweenness, global efficiency, clustering coefficient, and hub value.

SECONDARY OUTCOMES:
Change in Subjective Symptom Reporting | Days 1,2,3,4,5,6 through 7 inclusive post-injury
  Compare changes in daily cognitive and physical symptoms between the rest and exercise groups. Symptoms are rated on a 7 point Likert Scale.
Differences in Activity Levels | Days 1,2,3,4,5,6 through 7 inclusive post-injury
  Compare differences in activity levels between the rest and exercise groups. Activity levels are recorded by an accelerometer and will be compared to participant journal entries.

CONTACTS AND LOCATIONS:
Overall Officials: Naznin Virji-Babul, PhD, PT, Principal Investigator — Department of Physical Therapy, University of British Columbia
Locations (2):
- Canada (2):
  - Fortius Sport & Health, Burnaby, British Columbia
  - Djavad Mowafaghian Centre for Brain Health, Vancouver, British Columbia

REFERENCES:
- [Background] Thomas DG, Apps JN, Hoffmann RG, McCrea M, Hammeke T. Benefits of strict rest after acute concussion: a randomized controlled trial. Pediatrics. 2015 Feb;135(2):213-23. doi: 10.1542/peds.2014-0966. Epub 2015 Jan 5. PMID 25560444
- See also: Perception-Action Lab Website — http://pal.rehab.med.ubc.ca/
- See also: Fortius Sport & Health Website — http://www.fortiussport.com/Pages/default.aspx